CLINICAL TRIAL: NCT04830475
Title: Non-invasive Ventilation Prevents Post-operative Respiratory Failure in Patient Undergoing Bariatric Surgery
Brief Title: NIV Prevents Post-operative Respiratory Failure After Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Claudio Gambardella, Clinical Professor, University of Campania Luigi Vanvitelli
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NIV in obese
Record Dates: First submitted 2021-03-30; First posted 2021-04-05 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Obesity; Postoperative Respiratory Distress
MeSH Terms: conditions — Obesity | interventions — Noninvasive Ventilation

STUDY DESIGN:
Intervention Model Description: Retrospective Analysis
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NIV Group (Experimental): In poostoperative period, patients allocated in NIV Group fulfilled a 120-minute cycle of PSV + PEEP with full-face mask. Ventilation was performed with a Draeger Ventilator with the following basic settings: DeltaPInsp 10 mmHg + PEEP 5 mmHg + Fio2 60%.
  Interventions: Device: Non invasive ventilation (NIV)
- Control Group (Active Comparator): In the postoperative period, patients were offered VenturiMask with Fio2 60% at 15 l / m.
  Interventions: Device: Conventional Venturi Mask

INTERVENTIONS:
Device: Non invasive ventilation (NIV) — Patients allocated in NIV Group fulfilled a 120-minute cycle of PSV + PEEP with full-face mask. Ventilation was performed with a Draeger Ventilator with the following basic settings: DeltaPInsp 10 mmHg + PEEP 5 mmHg + Fio2 60%.
  Arms: NIV Group
Device: Conventional Venturi Mask — Patients were offered VenturiMask with Fio2 60% at 15 l / m.
  Arms: Control Group

SUMMARY:
Postoperative non-invasive ventilation (NIV) has been proposed as an attractive strategy to reduce morbidity and improve postoperative outcomes in obese subjects undergoing general anesthesia. Bariatric patients present a peculiar negative feature; the increased body mass index (BMI) correlates with loss of perioperative functional residual capacity (FRC), expiratory reserve volume (ERV) and total lung capacity (TLC), decreased up to 50% of preoperative values. The aim of the current randomized trial is to evaluate the efficacy of NIV in post-anaesthesia care unit (PACU) in reducing post-extubation acute respiratory failure and the consequent admission in intensive care units (ICU) after BIBP in obese adult patients.

ELIGIBILITY:
Inclusion Criteria:

* Morbid Obesity
* Patients undergoing Biliointestinal Bypass (BIBP)

Exclusion Criteria:

* Patients requiring emergency operation with rapid sequence induction
* Patients with suspected presence of difficult airway or pre-existing lung impairment
* Pregnancy
* Asthma
* Severe renal dysfunction,
* cardiac disease resulting in marked limitation of physical activity, corresponding to NYHA class >II

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-02-20 (Actual)

PRIMARY OUTCOMES:
Intensive care unit admission rate | 72 hours
  The primary outcome was the evaluation of the ICU admission rate after NIV in postoperative management of obese patients
Blood oxygen saturation (SaPo2) | 12 hours
  the evaluation of the oximetry values of obese patients after postoperative NIV adoption

CONTACTS AND LOCATIONS:
Locations (1):
- University of Campania Luigi Vanvitelli, Napoli, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Undecided